CLINICAL TRIAL: NCT04003272
Title: Post-market Clinical Follow-up Study to Provide Safety, Performance and Clinical Benefits Data of the Comprehensive Versa-Dial Reverse Titanium (Ti) Glenosphere in Primary, Fracture and Revision Total Shoulder Arthroplasty
Brief Title: MDR - Comprehensive Reverse/Versa Dial Ti Glenosphere
Status: Enrolling by invitation | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-40E
Record Dates: First submitted 2019-06-18; First posted 2019-07-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Shoulder Pain; Shoulder Injuries; Shoulder Fractures; Shoulder Arthritis; Shoulder Disease
MeSH Terms: conditions — Shoulder Pain; Shoulder Injuries; Shoulder Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Comprehensive Reverse Versa-Dial Titanium Glenosphere: Patients who have an allergy to typical cobalt chrome or other metal allergies had surgery to repair shoulder malfunction/disease.
  Interventions: Device: Comprehensive Reverse Versa-Dial Titanium Glenosphere

INTERVENTIONS:
Device: Comprehensive Reverse Versa-Dial Titanium Glenosphere — Implant used for patients with allergy to typical device material metals to repair shoulder malfunction/disease.

SUMMARY:
The objective of this retrospective/prospective consecutives series PMCF study is to collect data confirming safety, performance and clinical benefits of the Comprehensive Versa-Dial Reverse Ti Glenosphere when used for primary total shoulder arthroplasty (implants and instrumentation) at a 1,2,3,5,7, and 10- year follow-up* to meet EU Medical Device and other Regulatory Requirements for Post-Market Surveillance. Because Comprehensive Versa-Dial Reverse Ti Glenospheres have only been on the market since 2009, a prospective aspect to the study will be utilized as well to collect long-term data.

*The most recent available data will be used. If any of the listed time points are not available, data will be used from last available time point and follow-up will move forward at the closest available time point.

DETAILED DESCRIPTION:
The objective of this retrospective/prospective consecutives series PMCF study is to collect data confirming safety, performance and clinical benefits of the Comprehensive Versa-Dial Reverse Ti Glenosphere when used for primary total shoulder arthroplasty (implants and instrumentation) at a 1,2,3,5,7, and 10- year follow-up* to meet EU Medical Device and other Regulatory Requirements for Post-Market Surveillance. Because Comprehensive Versa-Dial Reverse Ti Glenospheres have only been on the market since 2009, a prospective aspect to the study will be utilized as well to collect long-term data.

The primary objective is the assessment of safety by analyzing implant survivorship. This will be established by recording the incidence and frequency of revisions, complications and adverse events. Relation of the events to either implant or instrumentation should be specified.

The secondary objective is the assessment of performance and clinical benefits by recording patient-reported clinical outcomes measures (PROMs).

*The most recent available data will be used. If any of the listed time points are not available, data will be used from last available time point and follow-up will move forward at the closest available time point.

ELIGIBILITY:
Inclusion Criteria:

* Biomet Comprehensive Reverse Shoulder products are indicated for use in patients whose shoulder joint has a grossly deficient rotator cuff with severe arthropathy and/or previously failed shoulder joint replacement with a grossly deficient rotator cuff. The patient must be anatomically and structurally suited to receive the implants and a functional deltoid muscle is necessary.

The Comprehensive Reverse Shoulder is indicated for primary, fracture, or revision total shoulder replacement for the relief of pain and significant disability due to gross rotator cuff deficiency.

Glenoid components with Hydroxyapatite (HA) coating applied over the porous coating are indicated only for uncemented biological fixation applications. The Glenoid Baseplate components are intended for cementless application with the addition of screw fixation.

Interlok™ finish humeral stems are intended for cemented use and the MacroBond™ coated humeral stems are intended for press-fit or cemented applications. Humeral components with porous coated surface coating are indicated for either cemented or uncemented biological fixation applications.

*** For the specific components, Titanium (Ti) Glenospheres are intended for patients with Cobalt Alloy material sensitivity.

Exclusion Criteria:

* Absolute contraindications include infection, sepsis, and osteomyelitis.

Relative contraindications include:

1. Uncooperative patient or patient with neurologic disorders who is incapable or unwilling to follow directions.
2. Osteoporosis.
3. Metabolic disorders which may impair bone formation.
4. Osteomalacia.
5. Distant foci of infections which may spread to the implant site.
6. Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram.
7. Patient is a prisoner.
8. Current alcohol or drug abuser.
9. If female, patient is known to be pregnant or breastfeeding.
10. Patient has a psychiatric illness or cognitive deficit that will not allow from proper informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive series of subjects implanted with the Comprehensive Versa-Dial Reverse Titanium (Ti) Glenosphere in primary, fracture and revision total shoulder arthroplasty according to the approved indications. Inclusion/exclusion criteria are identical to the indications and contraindications in the IFU.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2034-08-19 (Estimated); Study Completion 2035-09-01 (Estimated)

PRIMARY OUTCOMES:
Product Safety assessed through the incidence and frequency of revisions, complications and adverse events | Out to 10 years
  The primary objective is the assessment of safety by analyzing implant survivorship. This will be established by recording the incidence and frequency of revisions, complications, and adverse events. Relation of the events to either implant or instrumentation should be specified.

SECONDARY OUTCOMES:
Product Clinical Benefits and Performance evaluated through the Oxford Shoulder Scale OSS or Oxford Shoulder Questionnaire. | Out to10 years
  The secondary objective is the assessment of performance and clinical benefits by recording patient-reported clinical outcomes measures (PROMs) using the Oxford Shoulder Scale or Oxford Shoulder Questionnaire. The Scale ranges from 0-48 with 48 indicating a satisfactory joint function score. A score of 30-39 indicated moderate to mild arthritis, a score of 20-29 indicates moderate to severe arthritis and a score of 0-19 indicates severe arthritis.
Product Clinical Benefits and Performance evaluated through the Patient Assessment Questionnaire | Out to 10 years
  The secondary objective is the assessment of performance and clinical benefits by recording patient-reported clinical outcomes measures (PROMs). This will be accomplished through the use of the Patient Assessment Questionnaire where adverse events and/or complications (yes or no- if yes, an Adverse Event Report would be completed), patient's activity level with regard to operative side (wholly inactive, mostly inactive, sometimes participates in mild activities, regularly participates in mild activities, sometimes participates in moderate activities, regularly participates in moderate activities, regularly participates in active events, regularly participates in very active events, sometimes participates in impact sports, regularly participates in impact sports, or not recorded), and the Reported Score if Individual Scores are not available. (This would be the reported score of the Oxford Shoulder Scale as described above in Outcome 2).

CONTACTS AND LOCATIONS:
Overall Officials: Erin Osborn, Study Director — Zimmer Biomet
Locations (2):
- United States (2):
  - Norton Orthopaedic and Sports Medicine, Louisville, Kentucky
  - University of Buffalo, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No